CLINICAL TRIAL: NCT03670264
Title: BE Smokefree: Behavioral Economics Incentives to Engage Adolescents in Smoking Cessation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite efforts to recruit and enroll adolescents, identifying cigarette and e-cigarette users proved challenging. The study team was unable to meet the recruitment goal of 60 adolescents.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-014620; UL1TR001878 (NIH)
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quitline Incentive (Experimental): The incentive structure emphasizes engaging with the Quitline Delivered Treatment, with an additional smaller payment for tobacco cessation. Each adolescent can receive compensation for enrolling in the Quitline, for maintaining involvement in the Quitline program (per call for up to 5 calls), and, for those reporting abstinence, for submitting the cotinine swab and for confirmed quitting (negative salivary cotinine). Study procedures, payments and reminders are managed through the Way to Health (WTH) platform.
  Interventions: Behavioral: Quitline Incentive; Behavioral: Way to Health (WTH) Platform; Behavioral: Quitline Delivered Treatment
- Tobacco Cessation Incentive (Experimental): The incentive structure emphasizes quitting regardless of engagement with the Quitline Delivered Treatment (though the Quitline will be presented as a helpful tool). Each adolescent will receive compensation for enrolling in the Quitline and, for those reporting abstinence, compensation for submitting the cotinine swab and for confirmed quitting (negative salivary cotinine). Study procedures, payments and reminders are managed through the WTH platform.
  Interventions: Behavioral: Tobacco Cessation Incentive; Behavioral: Way to Health (WTH) Platform; Behavioral: Quitline Delivered Treatment
- No Financial Incentive (Placebo Comparator): No financial incentive to engage in Quitline Delivered Treatment or report abstinence. Study procedures and reminders are managed through the WTH platform.
  Interventions: Behavioral: Way to Health (WTH) Platform; Behavioral: Quitline Delivered Treatment

INTERVENTIONS:
Behavioral: Quitline Incentive — The incentive structure emphasizes engaging with the quitline, with an additional smaller payment for tobacco cessation. Each adolescent can receive compensation for enrolling in the quitline, for maintaining involvement in the quitline program (compensation per call for up to 5 calls), and, for those reporting abstinence, for submitting the cotinine swab and for confirmed quitting (negative cotinine swab).
  Arms: Quitline Incentive
Behavioral: Tobacco Cessation Incentive — The incentive payment structure emphasizes quitting regardless of engagement with the quitline (though the quitline will be presented as a helpful tool). Each adolescent will receive compensation for enrolling in the Quitline and, for those reporting abstinence, for submitting the cotinine swab and for confirmed quitting (negative cotinine swab).
  Arms: Tobacco Cessation Incentive
Behavioral: Way to Health (WTH) Platform — The WTH platform is a web-based platform that sends reminder text messages to participants regarding study procedures and has has secure financial tracking and processing systems to manage participant payments, including the ability to track earnings and pay participants via a non-integrated payment system.
Behavioral: Quitline Delivered Treatment — The quitline provides tobacco cessation treatment to individuals who enroll in treatment. This treatment includes 5 proactive counseling calls, each designed to help develop problem-solving and coping skills, secure social support, and plan for long-term abstinence. Participants can also call an 800 telephone number as needed for additional support between proactive calls.

SUMMARY:
More than 90% of adult smokers initiate tobacco use before age 18, making prevention and treatment of adolescent smoking a critical health priority. Behavioral economic interventions utilizing financial incentives can promote smoking cessation in adult populations. No studies have evaluated financial incentives among adolescents to promote engagement in effective tobacco cessation programs through primary care settings. The goal of this study is to to compare, through a pilot, randomized controlled trial, an intervention incentivizing contact with a tobacco cessation program (the Quitline), an intervention incentivizing quitting, or no financial incentive intervention on adolescent smoker enrollment and depth of engagement in the tobacco cessation program.

DETAILED DESCRIPTION:
Context:

Cigarette smoking remains a leading preventable cause of death in the United States (U.S.) with substantial morbidity, mortality, and financial costs each year. More than 90% of adult smokers initiate tobacco use before age 18, making prevention and treatment of adolescent tobacco use a critical health priority. Further, e-cigarettes are now the most common tobacco product used by teenagers, and adolescent use of e-cigarettes is strongly associated with transition to cigarette use. Behavioral economic interventions utilizing financial incentives can promote smoking cessation in adult populations. No studies have evaluated financial incentives among adolescents to promote engagement in effective tobacco cessation programs through primary care settings.

Objectives:

Primary Objective: To compare, through a pilot, randomized controlled trial, an intervention incentivizing contact with the Quitline, an intervention incentivizing quitting, or no financial incentive intervention on adolescent enrollment and depth of engagement in a tobacco cessation program (Free Smoker Quitline).

Secondary Objective: To compare cotinine-confirmed 2-month quit rates across the 3 groups, among users who report abstinence.

Study Design:

This is a randomized controlled trial of a Quitline incentive versus tobacco cessation incentive versus no financial incentive on adolescent engagement with a tobacco cessation program.

Setting/Participants:

Setting: Primary care sites within the Children's Hospital of Philadelphia (CHOP's) Pediatric Research Consortium along with other non-clinical community settings.

60 adolescent tobacco users will be recruited. Eligibility criteria include adolescents (aged 14-21 years), who speak English, screen positive for tobacco use during their routine well child or acute visit, are interested in quitting, and have a smart phone.

Study Interventions and Measures:

Adolescents will be randomized to 1 of 3 financial incentive groups: (1) Quitline Incentive: the payment structure emphasizes engaging with the Quitline, with an additional smaller payment for tobacco cessation; (2) Tobacco Cessation Incentive: the payment structure emphasizes quitting regardless of engagement with the quitline (though the quitline will be presented as a helpful tool); and (3) no financial incentive. The Quitline is funded by the Pennsylvania Department of Health and staffed by trained cessation counselors available 24 hours a day, 7 days a week.

Outcomes Measures: Objective 1: The main outcome of interest is adolescent completion of the tobacco cessation program, defined as the proportion of tobacco users identified in the clinic that enroll, use, and complete the Quitline program compared across the 3 groups. Objective 2: The secondary outcome is to confirm abstinence, via salivary cotinine concentration of <30 ng per milliliter at 10 weeks after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (aged 14-21 years), male or female, who speak English, screen positive for tobacco use (defined as having smoked cigarette(s) and/or used an e-cigarette product on at least 1 day during the 30 days before the clinical encounter) during their routine well child or acute visit, are interested in quitting, have a smart phone, and provide assent to participate.

Exclusion Criteria:

* Subjects that do not meet all of the inclusion criteria will not be enrolled.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jenssen, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Care Network, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quitline Incentive | Tobacco Cessation Incentive | No Financial Incentive
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quitline Incentive | Tobacco Cessation Incentive | No Financial Incentive | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.2 (1.6) | 16.6 (1.1) | 17.6 (2.1) | 17.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 4 | 2 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 5 | 5 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15
Number of participants enrolled in the Quitline [Count of Participants; unit: Participants] | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Program Completion
Description: Adolescent completion of the tobacco cessation program, defined as the proportion of tobacco users identified in the clinic that enroll, use, and complete the Quitline program compared across the 3 groups
Time Frame: 10 weeks
Population: The number of participants who enrolled in the Quitline
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline Incentive | Tobacco Cessation Incentive | No Financial Incentive
Number analyzed (Participants) | 5 | 5 | 5
Participants | 1 | 2 | 3

2. Secondary Outcome: Confirmation of Tobacco Abstinence
Description: Confirmation of abstinence will be measured by assessing if participants salivary cotinine concentration are <30 ng per milliliter
Time Frame: 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No adverse events occurred over the course of the study, of which each participant was enrolled in for 10 weeks.
Arm/Group | Quitline Incentive | Tobacco Cessation Incentive | No Financial Incentive
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
We were unable to reach our enrollment goal of 60 adolescents due to trouble recruiting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03670264/Prot_SAP_000.pdf